CLINICAL TRIAL: NCT06695923
Title: Association of Ultrafiltration Rates and Intradialytic Hypotension in Sohag University Hospitals.
Brief Title: Different Ultrafiltration Rates and Intradialytic Hypotension.
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Mahmoud Gad, Principal investigator and Resident in Internal medicine department, Sohag University Hospitals, Sohag University
Other Study IDs: Soh-Med--24-11-12MS
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-04

CONDITIONS: Hemodialysis; Intradialytic Hypotension
Keywords: Ultrafiltration rates; Intradialytic hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CBC Serum albumin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Finding relationship between different ultrafiltration rates and intradialytic hypotension in attempt to find the optimal cut off points.

DETAILED DESCRIPTION:
This observational study will be carried upon hemodialysis patients with different ultrafiltration rates at each session to study the association between ultrafiltration rates and intradialytic hypotension.

Thus identifying the optimal cut off of ultrafiltration rate points for each patient

ELIGIBILITY:
Inclusion Criteria:

All patients aged 18 Year or older on maintenance haemodialysis for at least 3 consecutive months receiving 3 sessions weekly.

-

Exclusion Criteria:

Patients aged < 18 years old.

Patients on recent haemodialysis < 3 months.

Pregnant women.

Patients with malignancy, severe infections or sepsis.

Patients with major bleeding.

Patients who cannot go upper limb monitoring of blood pressure.

Patients with severe heart failure (NYHA) class 3 or more.

Patients with severe anemia, Hemoglobin less than 6 g/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients more than 18 year old on maintenance hemodialysis receiving 3 sessions weekly.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Prevent intradialytic hypotension | 6 month
  Finding the optimal threshold of ultrafiltration rates to prevent intradialytic hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals,Faculty of medicine, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided